CLINICAL TRIAL: NCT00562744
Title: The Effect of High-Fidelity Simulation on Pediatric Advanced Life Support Training in Pediatric Housestaff: a Randomized Trial
Brief Title: Effect of Simulation on PALS Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Hospital of Philadelphia (Other)
Collaborators: Laerdal Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 2005-9-4379
Record Dates: First submitted 2007-11-21; First posted 2007-11-22 (Estimated); Last update posted 2007-11-22 (Estimated); Status verified 2007-11

CONDITIONS: Pediatric Housestaff

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SIM (Experimental): Participants complete training and assessment of performance in PALS scenarios using high-fidelity simulator
  Interventions: Other: Simulation
- MAN (No Intervention): Participants complete training and assessment of performance in PALS scenarios using mannequin

INTERVENTIONS:
Other: Simulation — Use of high-fidelity patient simulator for training and assessment of PALS scenario performance
  Arms: SIM

SUMMARY:
Patient simulation is a new and expanding technology that has proven effective as a teaching tool in various clinical settings, but data on pediatric simulation is lacking. Mock resuscitation scenarios have been shown in prior studies to be effective for improving knowledge, skill, and confidence in pediatric housestaff. Our objective is to assess the utility of a training program utilizing a human patient simulator of an infant as a teaching tool for pediatric housestaff training in resuscitation skills. We hypothesize that mock resuscitation exercises performed by pediatric housestaff on a patient simulator will result in improved performance on test scenarios when compared to the same training on a standard manikin.

DETAILED DESCRIPTION:
Patient simulation is a new and expanding technology that has proven effective as a teaching tool in various clinical settings, but data on pediatric simulation is lacking. Mock resuscitation scenarios have been shown in prior studies to be effective for improving knowledge, skill, and confidence in pediatric housestaff. Our objective is to assess the utility of a training program utilizing a human patient simulator of an infant as a teaching tool for pediatric housestaff training in resuscitation skills. We hypothesize that mock resuscitation exercises performed by pediatric housestaff on a patient simulator will result in improved performance on test scenarios when compared to the same training on a standard manikin.

We propose a randomized trial of pediatric residents of identical training levels from three children's hospitals. Participants will be assigned to a control group or an intervention group. The control group will undertake mock resuscitation scenarios on a standard manikin; the intervention group will perform the same exercises on a simulator. A test scenario will be administered at the end of each set of training scenarios and frequency and timing of a predetermined list of critical clinical assessments and interventions will be recorded. Analysis will consist of a comparison between control and intervention groups for success rates and time to completion for clinical assessments and interventions.

ELIGIBILITY:
Inclusion Criteria:

* PGY 1 or 2 in pediatrics at CHOP, St. Christopher's Hospital for Children, or A.I. DuPont Hospital for Children

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2006-01; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Cognitive performance in mock resuscitation scenarios | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Donoghue, MD, MSCE, Principal Investigator — CHOP
Locations (1):
- CHOP, Philadelphia, Pennsylvania, United States